CLINICAL TRIAL: NCT01845090
Title: Compared the Effect of Lanthanum Carbonate on Fibroblast Growth Factor 23 With Calcium Carbonate in Hemodialysis Patients
Brief Title: The Effect of Lanthanum Carbonate on Fibroblast Growth Factor 23
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Camillians Saint Mary's Hospital Luodong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SMHLANFGF23
Record Dates: First submitted 2013-04-24; First posted 2013-05-03 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2011-08

CONDITIONS: Other Nonspecific Abnormal Serum Enzyme Levels
MeSH Terms: interventions — lanthanum carbonate; Calcium Carbonate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lanthanum carbonate (Active Comparator): Lanthanum carbonate 375mg~750 mg tid for 6 months
  Interventions: Drug: Lanthanum carbonate
- Calcium carbonate (Active Comparator): Calcium carbonate 500mg~1000 mg tid for 6 months
  Interventions: Drug: Calcium Carbonate

INTERVENTIONS:
Drug: Lanthanum carbonate — the effect on serum FGF23
  Other Names: Fosrenol
  Arms: Lanthanum carbonate
Drug: Calcium Carbonate — Calcium carbonate 500mg~1000 mg tid for 6 months
  Other Names: TOP-CAL(CaCO3)
  Arms: Calcium carbonate

SUMMARY:
To compare the effect of lanthanum carbonate with calcium carbonate on serum FGF23 levels in hemodialysis patients.

DETAILED DESCRIPTION:
The investigators enrolled patients on maintenance hemodialysis and randomized them to two groups. One group will receive lanthanum carbonate and another group will receive calcium carbonate. The investigators will compare serum FGF23 levels between two groups after they receive above medication for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Chronic renal failure on maintenance hemodialysis 3 times a week for at least 3 months Serum calcium:8-10.5 mg/dL
* Serum phosphate:3.5-6 mg/dL(before washout period)
* Serum phosphate ≧6 mg/dL after washout period
* Serum i-PTH: 150-600 pg/mL

Exclusion Criteria:

* Diabetes mellitus
* Post parathyroidectomy
* Life expectancy< 6 months
* Liver disease(hepatitis B,C or liver dysfunction)
* Severe gastrointestinal disorders or other severe comorbidity
* Poor compliance
* Intolerance to lanthanum or calcium carbonate
* Active infection
* Malnutrition(serum albumin<3 g/dL or clinical assessment)
* Kt/V< 1.2 (inadequate dialysis)
* Serum phosphate>7.5 mg/dL after washout period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-08; Primary Completion 2014-07 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
serum level of fibroblast growth factor | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Shih-Ching Tsai, MD, Principal Investigator — Saint Mary's hospital-Lotung
Locations (1):
- Saint Mary's hospital-Lotung, Taipei, Taiwan

REFERENCES:
- [Derived] Natale P, Green SC, Ruospo M, Craig JC, Vecchio M, Elder GJ, Strippoli GF. Phosphate binders for preventing and treating chronic kidney disease-mineral and bone disorder (CKD-MBD). Cochrane Database Syst Rev. 2025 Jun 27;6(6):CD006023. doi: 10.1002/14651858.CD006023.pub4. PMID 40576086
- [Derived] Chang YM, Tsai SC, Shiao CC, Liou HH, Yang CL, Tung NY, Hsu KS, Chen IL, Liu MC, Kao JL, Jhen RN, Huang YT. Effects of lanthanum carbonate and calcium carbonate on fibroblast growth factor 23 and hepcidin levels in chronic hemodialysis patients. Clin Exp Nephrol. 2017 Oct;21(5):908-916. doi: 10.1007/s10157-016-1362-9. Epub 2016 Dec 7. PMID 27928636